CLINICAL TRIAL: NCT04152590
Title: Hospital-home Linkage Short-term Rehabilitation Therapy Using Real-time Interactive Digital Healthcare System in Post Operation Patients With Breast Cancer; Pilot Study
Brief Title: Real-time Interactive Digital Healthcare System in Post Operation Patients With Breast Cancer; Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JongIn Lee (Other)
Responsible Party: Sponsor-Investigator, JongIn Lee, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KC19EESI0325
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uincare (Experimental): Exercise using Uincare
  Interventions: Device: Uincare

INTERVENTIONS:
Device: Uincare — Interactive digital healthcare system

SUMMARY:
This study aims to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in post-operative patients with breast cancer. This is prospective pilot study. 20 breast cancer patients who underwent wide local excision-axillary lymph node diessection or modified radical mastectomy will be examined, and those with limited range of motion (ROM) of affected shoulder will be enrolled in the study. Shoulder ROM, Quick-DASH, pain evaluation with NRS, quality of life evaluation with FACT-B and EQ-5D will be evaluated on enrollment, 4-week, 8-week, and 12-weeks after enrollment.

DETAILED DESCRIPTION:
The limited range of motion (ROM) of the shoulder occur often after receiving breast cancer surgery, which may be due to post-operative pain, stiffness of shoulder girdle muscle, and etc. Due to this limited ROM, the patients may suffer difficulty in activities of daily life and quality of life may be reduced.

Uincare Homeplus is software manufactured in Korea, which uses infrared, kinect camera and motion capture technology to track 3D motion of the patients' articulation. Using this technology, the patients can receive feedback of their motion immediately.

The objective of the study is to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in post-operative patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent breast cancer surgery (wide local excision-axillary lymph node dissection or modified radical mastectomy)
* Limited active/passive range of motion of the affected shoulder (Flexion <160' or Abduction <160')
* post-operative day not exceeding 8 week
* Patients who agreed informed consent

Exclusion Criteria:

* Bilateral breast cancer surgery
* Patients with shoulder pain of limited ROM before breast cancer surgery
* Those unable to perform exercise due to general deconditioning
* Those with communication difficulty

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Range of motion of affected shoulder | Enrollment, 4 week, 8 week, 12 week
  Evaluation of change of range of motion of the affected shoulder from baseline to 12 weeks

SECONDARY OUTCOMES:
Numerical rating scale of affected shoulder | Enrollment, 4 week, 8 week, 12 week
  Evaluation of pain of the affected shoulder using numerical rating scale (0-10, with score 0 indicating no pain)
Functional outcome | Enrollment, 4 week, 8 week, 12 week
  Evaluation of shoulder function using Quick DASH
Quality of life of the patient with breast cancer | Enrollment, 4 week, 8 week, 12 week
  Evaluation of quality of life using FACT-B
Quality of life of the patient | Enrollment, 4 week, 8 week, 12 week
  Evaluation of quality of life using EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Jong In Lee, MD PhD, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, South Korea